CLINICAL TRIAL: NCT05785351
Title: Bariatric Surgery Benchmarks - How Much Do We Bench?
Brief Title: Swedish National Benchmarks in Laparoscopic Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Ebba Kihlstedt Pasquier, Principal Investigator, Region Östergötland
Other Study IDs: 2022-04311-01-1
Record Dates: First submitted 2023-01-06; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Bariatric Surgery
Keywords: Obesity; Bariatric Surgery; Laparoscopy; Benchmarking
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic Bariatric Surgery — Laparoscopic Bariatric Surgery: Gastric Sleeve and Roux-en-Y Gastric Bypass

SUMMARY:
The aim of this observational study is to define national reference values, according to the achievable benchmarks of care method (ABC™), for laparoscopic bariatric surgery in Sweden. The primary outcome is to identify the best possible, yet achievable, results during and after bariatric surgery. The second outcome to investigate if there are risk groups for complications, and if so perform risk-adjusted benchmark-calculations.

DETAILED DESCRIPTION:
The data source will be the Scandinavian Obesity Surgery Registry (SOReg), a prospective quality registry for obesity surgery. The time frame will be 2012-2021. The techniques to be investigated are laparoscopic roux-en-y gastric bypass and laparoscopic gastric sleeve respectively. Register variables related to surgical quality will be analyzed, and related to risk of peroperative and postoperative complications. The study will analyze data for the time of surgery and up to one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥ 18 years of age
* primary laparoscopic gastric sleeve or primary laparoscopic roux-en-y gastric bypass

Exclusion Criteria:

* other organ surgery at the time of the index operation
* no data about surgery
* no data about follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with obesity undergoing elective bariatric surgery in order to achieve weight loss.
Sampling Method: Probability Sample
Enrollment: 55372 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Benchmark values of variables related to surgical quality | Surgical intervention and up to one year after surgery
  ABC method of variables related to surgical quality (duration of surgery (minutes), complications (percentage), reoperations (percentage), weight loss at one year (percentage) etc)
Number of participants with severe postoperative complications | Within 30 days and one year after surgery
  Severe complication is defined as Clavien-Dindo grade ≥ IIIa

SECONDARY OUTCOMES:
Potential risk groups for complications | Within 30 days and one year after surgery
  Estimated with multivariable regression analysis looking at BMI (kg/m^2), age categories, gender, waist line category, occurrence of dyspepsia, hypertension, previous thrombo-embolism or diabetes
Risk-adjusted benchmark values | Within 30 days and one year after surgery
  ABC method of any identified risk group(s) for complications

IPD SHARING:
Plan to Share IPD: No